CLINICAL TRIAL: NCT00002400
Title: An Open-Label Randomized Study of Delavirdine Mesylate (Rescriptor) in Combination With Zidovudine (Retrovir) and Two Doses of Indinavir (Crixivan) Versus Zidovudine, Lamivudine (Epivir), and Indinavir in HIV-1-Infected Individuals
Brief Title: A Study of Two Anti-HIV Drug Combinations in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmacia and Upjohn (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 228C; 0063
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-01

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; Indinavir; RNA, Viral; Delavirdine; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Delavirdine; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Delavirdine mesylate
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of giving HIV-infected patients delavirdine (DLV) plus zidovudine (ZDV) plus 2 doses of indinavir (IDV) or ZDV plus IDV plus lamivudine (3TC). This study also examines how the body processes DLV when it is given in combination with other drugs.

DETAILED DESCRIPTION:
In this multicenter, open-label study, 45 HIV-1-positive patients receive either combination drug therapy with delavirdine (DLV), zidovudine (ZDV), and indinavir (IDV) or combination drug therapy with ZDV, lamivudine (3TC), and IDV. NOTE: Patients are treated for 24 weeks and may opt to continue on study for 24 additional weeks, if HIV-1 RNA is less than 5,000 copies/ml or at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 positive.
* CD4 count above 50.
* HIV-1 RNA greater than 20,000.

Prior Medication:

Allowed:

Less than 1 month prior treatment with zidovudine.

Exclusion Criteria

Prior Medication:

Excluded:

* Prior 3TC, protease inhibitors, or non-nucleoside reverse transcriptase inhibitors.
* Prior ZDV of greater than 1 month total duration.

Prior Treatment:

Excluded:

* Lamivudine.
* Protease inhibitors.
* Non-nucleoside reverse transcriptase inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacia & Upjohn, Peapack, New Jersey, United States